CLINICAL TRIAL: NCT03522714
Title: A Prospective, Randomized Controlled Trial Evaluating the Effectiveness of the Fluid Immersion Simulation (FIS) System Versus Air Fluidized Bed (AFB) System in the Acute Post-Operative Management of Surgically Closed Pressure Ulcers
Brief Title: Fluid Immersion Simulation (FIS) System Versus Air Fluidized Bed (AFB) System for Pressure Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Robert Galiano, Associate Professor of Surgery (Plastic Surgery) and Dermatology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU00200584
Record Dates: First submitted 2018-02-13; First posted 2018-05-11 (Actual); Results first posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Pressure Ulcer
Keywords: support; flap; pressure; surface; closure; ulcer
MeSH Terms: conditions — Pressure Ulcer; Ulcer

STUDY DESIGN:
Intervention Model Description: 1:1 allocation ratio
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Fluid Immersion Simulation System (FIS) (Active Comparator): Pressure ulcer patients are assigned to Fluid Immersion Simulation System (Dolphin) after operative debridement and closure.
  Interventions: Device: Fluid Immersion Simulation System
- Air Fluidized Bed System (AFB) (Active Comparator): Pressure ulcer patients are assigned to Air Fluidized Bed (Clinitron) after operative debridement and closure
  Interventions: Device: Air Fluidized Bed System

INTERVENTIONS:
Device: Fluid Immersion Simulation System — Dolphin Fluid Immersion Simulation® System Mattress will be used
  Other Names: FIS, Dolphin
  Arms: Fluid Immersion Simulation System (FIS)
Device: Air Fluidized Bed System — Air Fluidized Bed (Clinitron) will be used.
  Other Names: AFB, Clinitron
  Arms: Air Fluidized Bed System (AFB)

SUMMARY:
The primary objective is to compare the efficacy of the FIS on closure rate to the AFB after 2 weeks of operative debridement and closure.

DETAILED DESCRIPTION:
Secondary Objectives:

1. Compare the complication rate in each treatment group during the acute postoperative period (2 weeks).
2. Comparisons of the inflammatory and bacterial microbiomes of pressure ulcers following surgical therapy.
3. Comparisons of baseline patient characteristics and their relationship to both early and late pressure ulcer recurrence, and complication rates.
4. Assessment of outcomes and complications associated with flap technique and surgeon guided descriptions of the operative closure.
5. Compare the absolute costs associated with the FIS System against AFB system.
6. Compare the acceptance of each system by subjects and nursing staff, including the parameter of patient comfort at 7 and 14 days postoperative.
7. Assessing the incidence of complications and additional treatments needed following the two week study period.

ELIGIBILITY:
Inclusion Criteria:

1. will be admitted as an inpatient
2. is ≥ 18 years of age and ≤ 85 years of age at time of consent
3. is able to provide his/her own informed consent
4. is deemed by the investigators to be reasonably compliant
5. has a pressure ulcer meeting criteria for stage III or IV
6. has not participated in a clinical trial within the past 30 days
7. has a 30-day wound history available if the wound has been previously treated

Exclusion Criteria:

1. has a life expectancy of < 12 months
2. is not healthy enough to undergo surgery for any reason
3. has a history of radiation therapy
4. is, in the opinion of the investigator, noncompliant
5. has a history of > 3 closures of pressure ulcers in the same site
6. has a history of a bleeding disorder
7. has severe fecal incontinence

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-08-08 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert D Galiano, MD, Principal Investigator — Northwestern Medicine
Locations (1):
- Northwestern Memorial Hospital Plastic Surgery, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fluid Immersion Simulation System (FIS) | Air Fluidized Bed System (AFB)
Started | 38 | 42
Completed | 28 | 40
Not Completed | 10 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluid Immersion Simulation System (FIS) | Air Fluidized Bed System (AFB) | Total
Number analyzed (Participants) | 38 | 42 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 42 | 80
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.61 (13.75) | 47.45 (42) | 48.48 (13.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 12 | 27
  Male | 23 | 30 | 53
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic | 1 | 6 | 7
  White | 27 | 20 | 47
  African American | 10 | 15 | 25
  Other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 38 | 42 | 80

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Successful Closure of Wound at 2 Weeks After Surgery
Description: Comparison of success of closure between treatment groups.
Time Frame: 2 weeks
Measure: Number; unit: percent of participants
Arm/Group | Fluid Immersion Simulation System (FIS) | Air Fluidized Bed System (AFB)
Number analyzed (Participants) | 28 | 40
percent of participants | 85.7142857 | 87.5

2. Secondary Outcome: Number of Participants With Complications
Description: Comparison of complication rate, including dehiscence, necrosis, maceration, and seromas between treatment groups. These are gathered via the patient's medical chart and interaction with the Principle Investigator (their physician).
Time Frame: 2 weeks
Measure: Number; unit: Participants
Arm/Group | Fluid Immersion Simulation System (FIS) | Air Fluidized Bed System (AFB)
Number analyzed (Participants) | 28 | 40
Participants
  Complications Prior to ClimateCare introduction | 8 | 15
  Complications Following ClimateCare introduction | 17 | 20

3. Secondary Outcome: Differences in Quantitative Patient Survey Responses: Acceptability
Description: Differences in quantitative patient survey responses regarding acceptability. This scale includes three subscales: 1) comfort, 2) difficulty with mobilization, and 3) pain at surgical site. Each subscale is graded on a scale of 1-5 with 1 being "better" (i.e. very comfortable, no difficulty, or no pain) and 5 being "worse" (i.e. very uncomfortable, extreme difficulty, or extreme pain). Subscales will be combined to compute a total score by averaging the sum of each of the three subscales. The total score indicates patient acceptability on a scale of 1-5 with 1 being "better" (very acceptable) and 5 being "worse" (not acceptable).
Time Frame: 2 weeks
Measure: Mean (Full Range); unit: Scores on a scale
Arm/Group | Fluid Immersion Simulation System (FIS) | Air Fluidized Bed System (AFB)
Number analyzed (Participants) | 28 | 40
Scores on a scale | 2.08 [1 to 5] | 2.06 [1 to 5]

4. Secondary Outcome: Differences in Quantitative Nurse Survey Responses
Description: Differences in quantitative nurse survey responses regarding acceptability and tolerance of each therapeutic modality, including patient comfort. This survey includes three subscales: 1) ease of use, 2) amount of training required, and 3) Time Required for Troubleshooting or Otherwise Occupied by Device. Each subscale is graded on a scale of 1-5 with 1 being "better" (i.e. no difficulty, no training, or no time) and 5 being "worse" (i.e. extreme difficulty, very high amount of training, or >30 minutes a day). Subscales will be combined to compute a total score by averaging the sum of each of the three subscales. The total score indicates nurse acceptability on a scale of 1-5 with 1 being "better" (very acceptable) and 5 being "worse" (not acceptable).
Time Frame: 2 weeks
Measure: Mean (Full Range); unit: Scores on a scale
Arm/Group | Fluid Immersion Simulation System (FIS) | Air Fluidized Bed System (AFB)
Number analyzed (Participants) | 28 | 40
Scores on a scale | 1.49 [1 to 5] | 1.72 [1 to 5]

ADVERSE EVENTS:
Time Frame: Baseline to 1 year.
Arm/Group | Fluid Immersion Simulation System (FIS) | Air Fluidized Bed System (AFB)
All-Cause Mortality (participants affected / at risk) | 4/38 | 2/42
Serious Adverse Events (participants affected / at risk) | 0/38 | 1/42
Other Adverse Events (participants affected / at risk) | 22/38 | 10/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fluid Immersion Simulation System (FIS) (N=38) | Air Fluidized Bed System (AFB) (N=42)
Severe Dehiscence (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fluid Immersion Simulation System (FIS) (N=38) | Air Fluidized Bed System (AFB) (N=42)
Minor Complications (Skin and subcutaneous tissue disorders) | 22 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-20): https://cdn.clinicaltrials.gov/large-docs/14/NCT03522714/Prot_SAP_000.pdf
  • Informed Consent Form (2019-06-28): https://cdn.clinicaltrials.gov/large-docs/14/NCT03522714/ICF_001.pdf